CLINICAL TRIAL: NCT04700956
Title: Does Prophylactic Mesh Placement in Emergency Midline Laparotomy Reduce the Incidence of Incisional Hernia? A Prospective Randomized Clinical Trial
Brief Title: Does the Use of Prophylactic Mesh Reduce Incisional Hernia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Eşref Ulutaş, Research assistant, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20202020
Record Dates: First submitted 2020-12-19; First posted 2021-01-08 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Incisional Hernia
Keywords: incisional hernia; prophylactic; mesh; emergency surgery
MeSH Terms: conditions — Incisional Hernia | interventions — Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the primary suture group (Active Comparator): The linea alba will be closed to a ratio of 5mm / 5mm. Only the fascia will be sutured ; fat or muscle tissue will be avoided. Subcutaneous tissue will be closed with polyglactin 3/0 suture. The skin will be closed with a stapler.
  Interventions: Procedure: primary abdominal closure
- mesh group (Experimental): After the fascia was closed with the same method, 5 cm of subcutaneous tissue will be dissected around the incision. The mesh will be placed in the supra-aponeurotic area (onlay) to a distance of laterally and cranial-caudally 5 cm from the fascia margins. The mesh used will be partially absorbable, light and large porous. After this procedure, the borders of the mesh will be fixed circumferentially on the abdominal wall using polypropylene suture to prevent the intestines from herniating on the mesh. Two subcutaneous drainage catheters will be placed in all patients with mesh.
  Interventions: Device: abdominal closure with prophylactic mesh

INTERVENTIONS:
Procedure: primary abdominal closure — The linea alba will be closed to a ratio of 5mm / 5mm. Only the fascia will be sutured ; fat or muscle tissue will be avoided. Subcutaneous tissue will be closed with polyglactin 3/0 suture. The skin will be closed with a stapler.
  Other Names: primary abdominal closure with suture
  Arms: the primary suture group
Device: abdominal closure with prophylactic mesh — After the fascia was closed with the same method, 5 cm of subcutaneous tissue will be dissected around the incision. The mesh will be placed in the supra-aponeurotic area (onlay) to a distance of laterally and cranial-caudally 5 cm from the fascia margins. The mesh used will be partially absorbable, light and large porous. After this procedure, the borders of the mesh will be fixed circumferentially on the abdominal wall using polypropylene suture to prevent the intestines from herniating on the mesh. Two subcutaneous drainage catheters will be placed in all patients with mesh.
  Arms: mesh group

SUMMARY:
Incisional hernia is a common condition after abdominal surgery. Because linea alba has less vascularity, incisional hernia more common in midline incisions. It is seen in the general population between 11-20%. In some high-risk situations, this rate increases up to 40-69% (abdominal aortic aneurysm, morbid obesity, colorectal surgery).It is known that incisional hernia that occurs in the postoperative period can lead to emergency surgical causes such as incarceration-strangulation, has a significant share in health expenses and seriously impairs the quality of life in patients.One of the methods tried to reduce incisional hernia is the use of mesh. But this abdominal closure technique is not used routinely in our country and the other countries. This study will be important of the studies in Turkey and world for patient selection in prophylactic mesh use, techniques to be applied and early / late results.

The aim of the study is to compare the classical abdominal closure technique with use of mesh in order to minimize the incisional hernia and associated complications after midline laparotomy.

DETAILED DESCRIPTION:
Background

There are patient and surgical procedure-related risk factors that increase the risk of postoperative incisional hernia. Patient-related risk factors: male gender, previous laparotomy, over 50 years of age, malignant disease, COPD, hypoalbuminemia, sepsis, obesity (BMI> 30 kg / m2), anemia, DM, used to steroid, smoking, chemoterapi, cardiovascular disease, RT to the abdominal wall and to be postoperative abdominal wall defects. In studies conducted in many centers around the world, it has been shown that the use of prophylactic mesh reduces the incidence of incisional hernia, especially in high-risk patients. When the literature was reviewed, reviews and meta-analyzes about the use of prophylactic mesh showed a significant decrease in incisional hernia incidence. However, routine practice has not yet been recommended, as long-term follow-up results and secondary results (complications, cost analysis, quality of life) are not clearly explained. However, it has been reported that higher quality studies are needed.

This abdominal closure technique is not used routinely in our country. This study will be one of the first studies in Turkey for patient selection in prophylactic mesh use, techniques to be applied and early / late results.

The aim of the study is to compare the classical abdominal closure technique with use of mesh in order to minimize the incisional hernia and associated complications after midline laparotomy.

Method

Patients aged 18 years and over who were scheduled to undergo emergency abdominal surgery with midline laparotomy will be randomly assigned (1: 1) to primary abdominal closure or mesh group via a computer-generated randomization sequence.

Detailed information was given to all patients before they were included in the study, and their informed consent forms were recorded.

The method in the primary suture group: The linea alba will be closed to a ratio of 5mm / 5mm. Only the fascia will be sutured ; fat or muscle tissue will be avoided. Subcutaneous tissue will be closed with polyglactin 3/0 suture. The skin will be closed with a stapler.

Method in the mesh group: After the fascia was closed with the same method, 5 cm of subcutaneous tissue will be dissected around the incision. The mesh will be placed in the supra-aponeurotic area (onlay) to a distance of laterally and cranial-caudally 5 cm from the fascia margins. The mesh used will be partially absorbable, light and large porous. After this procedure, the borders of the mesh will be fixed circumferentially on the abdominal wall using polypropylene suture to prevent the intestines from herniating on the mesh. Two subcutaneous drainage catheters will be placed in all patients with mesh.

Antithrombotic prophylaxis with low molecular weight heparin, antibiotic prophylaxis with cefazolin and metronidazole will be applied to all patients according to the hospital protocol.

Power analysis; To provide sufficient statistical power, sample size calculation was made. Incisional hernia rates were estimated between 5% and 25% between the two groups. It was calculated that 49 patients per group with 80% test power in the 95% confidence interval would be needed. In the follow-up period, it was planned to include 52 patients in each group, with the prediction that 5% of the patients would be excluded from the study.

Data Entry and Statistical Analysis; Kolmogorov-Smirnov and Shapiro-Wilk normality tests will be carried out before starting the statistical analysis. If normality cannot be achieved even in one of the groups, non-parametric test methods will be selected. Next, the Mann-Whitney U test will be used to compare the variables obtained by the measurement between the two groups.

Chi-square and Fisher Final tests will be used to analyze the relationships or differences between groups in terms of categorical variables.

Univariate logistic regression analysis will be performed to determine the factors thought to cause an incisional hernia. Then, multivariate logistic regression analysis will be done for variables with

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18 years of age,
* laparotomy with the midline incision of the abdomen,
* all emergency surgery indications,
* having at least two of the risk factors.

Exclusion Criteria:

* Patients under 18 years of age,
* elective surgeries,
* off-midline incisions,
* concurrent hernia,
* laparoscopic surgery,
* history of metastatic cancer,
* life expectancy less than 2 years,
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-12-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
primary outcome | up to one year
  incisional hernia rate

SECONDARY OUTCOMES:
secondary outcome | up to one months
  seroma rate
secondary outcome | up to one months
  hematoma rate
secondary outcome | up to ten days
  burst abdomen rate
secondary outcome | up to one months
  deep vein thymbosis rate
secondary outcome | up to one months
  pulmonary and cardiac complication rate
secondary outcome | up to one hundred twenty minutes
  mean operation time (minute)
secondary outcome | up to twenty days
  mean hospital stay time (day)
secondary outcome | up to one year
  chronic pain rate (visual analog scale, VAS)
secondary outcome | up to one year
  quality of life measures (0-100 points) - It will be measured using the EQ-5D test.
secondary outcome | up to one year
  re-operation rate

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University Konya City Hospital General Surgery Department, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jairam AP, Lopez-Cano M, Garcia-Alamino JM, Pereira JA, Timmermans L, Jeekel J, Lange J, Muysoms F. Prevention of incisional hernia after midline laparotomy with prophylactic mesh reinforcement: a meta-analysis and trial sequential analysis. BJS Open. 2020 Jun;4(3):357-368. doi: 10.1002/bjs5.50261. Epub 2020 Feb 14. PMID 32057193
- [Result] Argudo N, Iskra MP, Pera M, Sancho JJ, Grande L, Lopez-Cano M, Pereira JA. The use of an algorithm for prophylactic mesh use in high risk patients reduces the incidence of incisional hernia following laparotomy for colorectal cancer resection. Cir Esp. 2017 Apr;95(4):222-228. doi: 10.1016/j.ciresp.2017.03.010. Epub 2017 Apr 8. English, Spanish. PMID 28400141
- [Result] Bhangu A, Fitzgerald JE, Singh P, Battersby N, Marriott P, Pinkney T. Systematic review and meta-analysis of prophylactic mesh placement for prevention of incisional hernia following midline laparotomy. Hernia. 2013 Aug;17(4):445-55. doi: 10.1007/s10029-013-1119-2. Epub 2013 May 28. PMID 23712289
- [Result] Fischer JP, Basta MN, Wink JD, Krishnan NM, Kovach SJ. Cost-utility analysis of the use of prophylactic mesh augmentation compared with primary fascial suture repair in patients at high risk for incisional hernia. Surgery. 2015 Sep;158(3):700-11. doi: 10.1016/j.surg.2015.02.030. Epub 2015 Jul 15. PMID 26189071
- [Result] Kurmann A, Barnetta C, Candinas D, Beldi G. Implantation of prophylactic nonabsorbable intraperitoneal mesh in patients with peritonitis is safe and feasible. World J Surg. 2013 Jul;37(7):1656-60. doi: 10.1007/s00268-013-2019-4. PMID 23568247
- [Result] Llaguna OH, Avgerinos DV, Nagda P, Elfant D, Leitman IM, Goodman E. Does prophylactic biologic mesh placement protect against the development of incisional hernia in high-risk patients? World J Surg. 2011 Jul;35(7):1651-5. doi: 10.1007/s00268-011-1131-6. PMID 21547421
- [Result] Payne R, Aldwinckle J, Ward S. Meta-analysis of randomised trials comparing the use of prophylactic mesh to standard midline closure in the reduction of incisional herniae. Hernia. 2017 Dec;21(6):843-853. doi: 10.1007/s10029-017-1653-4. Epub 2017 Sep 1. PMID 28864937
- [Result] San Miguel C, Melero D, Jimenez E, Lopez P, Robin A, Blazquez LA, Lopez-Monclus J, Gonzalez E, Jimenez C, Garcia-Urena MA. Long-term outcomes after prophylactic use of onlay mesh in midline laparotomy. Hernia. 2018 Dec;22(6):1113-1122. doi: 10.1007/s10029-018-1833-x. Epub 2018 Oct 4. PMID 30288617
- [Result] Garcia-Urena MA, Lopez-Monclus J, Hernando LA, Montes DM, Valle de Lersundi AR, Pavon CC, Ceinos CJ, Quindos PL. Randomized controlled trial of the use of a large-pore polypropylene mesh to prevent incisional hernia in colorectal surgery. Ann Surg. 2015 May;261(5):876-81. doi: 10.1097/SLA.0000000000001116. PMID 25575254